CLINICAL TRIAL: NCT03923283
Title: End-tidal Carbondioxide Levels Under Surgery Drapes During Local Eye Surgery: Retrospective Study
Brief Title: The Measurements of End-tidal Carbondioxide Levels
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Ilknur Suidiye, Assistant Professor, Duzce University
Other Study IDs: Duzce University
Record Dates: First submitted 2017-06-05; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Other Disorders of the Eye Following Cataract Surgery
Keywords: End-tidal carbondioxide; surgery drapes; carbondioxide accumulation; eye surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose: The aim of this retrospective study is to investigate the end tidal carbon dioxide pressure (ETCO2) values in order to determine the carbon dioxide accumulation under drape and to investigate it's hemodynamic effects based on anesthetic and surgical records in eye surgeries under local anesthesia.

Methods: The data were collected from anesthetic records of the patients who were followed with noninvasive capnograph (Capnostream 20 p, Oridion®, Israel) by the anesthesiology department in the operating room at Duzce University Faculty of Medicine Hospital during the period of January 2016 to December 2016.

Collected data from the 42 patients' records were systolic, diastolic and mean arterial pressures, operation duration, total local anesthetic and, heart rate, ST segment analysis, ETCO2 pressure, pulse oximeter values.

The time periods of collected datas were determined as: after the anesthesia and before drape closure (baseline level), at 10th, 15th, 20th, 45th of the surgery and 5 minutes after drape removal.

DETAILED DESCRIPTION:
After approval from the Duzce Faculty of Medicine Noninvasive Researches Ethics Committee (02.01.2017), the datas were collected patients anesthetic forms who were followed with capnograph (Capnostream 20 p, Oridion, Israel) by the anesthesiology department for eye surgery in the operating room at Duzce University Faculty of Medicine Hospital during the period of 01 January 2016 to 31 December 2016. It was observed that 42 patient records met the study criteria. Demographic and clinical datas were abstracted from anesthetic and clinical records.

Age, weight, height of the patients, operation types, operation duration times, local anesthetic performing types, noninvasive systolic, diastolic and mean arterial pressures, cardiac rates, ST segment analysis (Datex Ohmeda monitor, GE Health Care, Finland) ( This monitor use for the routine monitorisation in the eye surgery operating room in our hospital) systolic, diastolic and mean arterial pressure measurements, end tidal carbon dioxide levels, pulse oximeter values were extracted from anesthetic forms retrospectively.

Arrhythmia recordings were evaluated as (yes / no) over time periods. Surgical field was covered with reusable cotton fabric drape or dispossible surgical adhesive plastic drape (SteriDrape, 3M). We included the patients records who were covered with the same kind of drapes (SteriDrape, 3M). We excluded records with another type of drapes usage or without any data about drape type to provide the homogenisation and clearity of the results.

Datas were collected from the anesthetic forms which time periods were determined as the baseline, before closing drape, at 10th, 15th, 20th, 45th minutes after covering and 5 minutes after drape removal. Records with pulmonary disease, diabetes mellitus and sedative usage, alcohol usage were excluded from the study.

The comparisons were made with patients basal status and time periods statistically.

ELIGIBILITY:
Inclusion Criteria:

* Datas were collected after approval from the Duzce Faculty of Medicine Noninvasive Researches Ethics Committee (02.01.2017), the datas of the patients who were followed with capnograph (Capnostream 20 p, Oridion, Israel) by the anesthesiology departhment in the operating room at Duzce University Faculty of Medicine hospital during the period of January 2016 to December 2016 .

Exclusion Criteria:

* Patients with chronic obstructive pulmonary disease, diabetes mellitus and sedative usage were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients who were followed with capnograph (Capnostream 20 p, Oridion, Israel) by the anesthesiology departhment in the operating room at Duzce University Faculty of Medicine hospital during the period of January 2016 to December 2016 was collected.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
The Measurements of End-tidal Carbondioxide Levels Under Surgery Drapes During Local Eye Surgery | 1 hour
  To determine the difference between capnostream capnography and carbon dioxide levels measured at various times in patients undergoing eye surgery under local anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Ilknur S Yorulmaz, Principal Investigator — Duzce University Faculty Of Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dinsmore M, Han JS, Fisher JA, Chan VW, Venkatraghavan L. Effects of acute controlled changes in end-tidal carbon dioxide on the diameter of the optic nerve sheath: a transorbital ultrasonographic study in healthy volunteers. Anaesthesia. 2017 May;72(5):618-623. doi: 10.1111/anae.13784. Epub 2017 Feb 8. PMID 28177116
- [Background] Allen JG, MacNaughton P, Satish U, Santanam S, Vallarino J, Spengler JD. Associations of Cognitive Function Scores with Carbon Dioxide, Ventilation, and Volatile Organic Compound Exposures in Office Workers: A Controlled Exposure Study of Green and Conventional Office Environments. Environ Health Perspect. 2016 Jun;124(6):805-12. doi: 10.1289/ehp.1510037. Epub 2015 Oct 26. PMID 26502459
- [Background] Howarth C, Sutherland B, Choi HB, Martin C, Lind BL, Khennouf L, LeDue JM, Pakan JM, Ko RW, Ellis-Davies G, Lauritzen M, Sibson NR, Buchan AM, MacVicar BA. A Critical Role for Astrocytes in Hypercapnic Vasodilation in Brain. J Neurosci. 2017 Mar 1;37(9):2403-2414. doi: 10.1523/JNEUROSCI.0005-16.2016. Epub 2017 Jan 30. PMID 28137973
- [Background] Weeke LC, Dix LML, Groenendaal F, Lemmers PMA, Dijkman KP, Andriessen P, de Vries LS, Toet MC. Severe hypercapnia causes reversible depression of aEEG background activity in neonates: an observational study. Arch Dis Child Fetal Neonatal Ed. 2017 Sep;102(5):F383-F388. doi: 10.1136/archdischild-2016-311770. Epub 2017 Jan 27. PMID 28130246
- [Background] Courtney P. The National Cataract Surgery Survey: I. Method and descriptive features. Eye (Lond). 1992;6 ( Pt 5):487-92. doi: 10.1038/eye.1992.103. PMID 1286712
- [Background] Report of the Joint Working Party on anesthesia in Ophthalmic Surgery. Royal Collage of Anaesthetists and Collage of Ophthalmologists, March (1993).
- [Background] Jerusalem E, Starling EH. On the significance of carbon dioxide for the heart beat. J Physiol. 1910 May 13;40(4):279-94. doi: 10.1113/jphysiol.1910.sp001370. No abstract available. PMID 16993008